CLINICAL TRIAL: NCT01794364
Title: A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo-Controlled, Single Dose Escalating Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-06291874 After Administration Under Fasted And Fed Conditions In Healthy Adult Subjects
Brief Title: Single Dose Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Study Of PF-06291874 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B4801009
Record Dates: First submitted 2012-12-21; First posted 2013-02-18 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: T2DM; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-06291874

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: Cohort A (Experimental): Each subjects in Cohort A will receive 2 single doses of PF-06291874 and 1 placebo dose in random order in Periods 1-3; in addition, 1 dose of PF-06291874 will be administered in Period 4 in the fed state.
  Interventions: Drug: PF-06291874; Other: placebo

INTERVENTIONS:
Drug: PF-06291874 — PF-06291874 will be administered as an extemporaneously prepared suspension for all doses within the initially planned range of 75 mg to 500 mg.
Other: placebo — Correspondingly, placebo doses will be administered as suspension.

SUMMARY:
The primary purpose of this trial is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of single oral doses of PF-06291874 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including clinically significant drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0-72/dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] | 0-72/dose
Maximum Observed Plasma Concentration (Cmax) | 0-72/dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-72/dose
Plasma Decay Half-Life (t1/2) | 0-72/dose
Apparent Oral Clearance (CL/F) | 0-72/dose
Apparent Volume of Distribution (Vz/F) | 0-72/dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4801009&StudyName=Single%20Dose%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Study%20Of%20PF-06291874%20In%20Healthy%20Adult%20Subjects%20